CLINICAL TRIAL: NCT01353235
Title: A Prospective Randomized Trial of Systemic Corticosteroids (Oral Prednisolone) in Severe Exacerbation of COPD Requiring Ventilatory Assistance
Brief Title: Oral Prednisolone in Severe Acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fekri Abroug (Other)
Responsible Party: Sponsor-Investigator, Fekri Abroug, ead of the ICU, Hôpital Universitaire Fattouma Bourguiba
Organization: Hôpital Universitaire Fattouma Bourguiba (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: steroids in COPD exacerbation
Record Dates: First submitted 2011-05-10; First posted 2011-05-13 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: COPD Exacerbation
Keywords: COPD; acute respiratory failure; mechanical ventilation; non invasive ventilation; steroids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (Sham Comparator)
  Interventions: Drug: usual care
- Prednisolone (Active Comparator): 1mg/kg/day prednisolone for the entire ICU stay and a maximum of 10 days
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Patients assigned to corticotherapy arm, will receive oral prednisolone 1mg/kg/j as an add on therapy for a maximum of 10 days.
  Arms: Prednisolone
Drug: usual care — no drug administered
  Arms: usual care

SUMMARY:
Evaluation of systematic administration of oral prednisolone (1mg/Kg/day) as an add on therapy in Chronic Obstructive Pulmonary Disease (COPD) patients admitted to intensive care unit (ICU) for severe exacerbation of COPD. Patients with pneumonia are excluded.

Randomization is stratified according to ventilatory support: non invasive or conventional ventilation.The major outcome is the ICU mortality rate in overall population and stratified according to ventilatory mode (noninvasive ventilation (NIV) versus conventional).

Secondary outcomes are superinfection necessitating a new antibiotic course, Length of mechanical ventilation (MV) (and ventilatory free days), Length of ICU stay, The frequency of gastric bleeding episodes that of frequency of hyperglycemic episodes.

ELIGIBILITY:
Inclusion Criteria:

* All COPD patients (according to the ATS definition) experiencing acute exacerbation originating in acute respiratory failure and requiring ICU admission will be included in the study.

COPD exacerbation is defined by the increased frequency of cough, volume and purulence of sputum and that of wheeze.

Acute respiratory failure is defined by the presence of hypercapnia with PaCO2 >45mmHg associated with pH > 7.35 and signs of respiratory muscle fatigue (contraction of accessory respiratory muscles, thoracoabdominal swinging ,..).

Exclusion Criteria:

* Asthmatic patients defined by a reversible obstructive disease following nebulized bronchodilators,
* Patients with uncontrolled left heart failure,
* AECOPD patients with a radiologically documented pneumonia,
* Systemic corticotherapy within 30 days before screening,
* contra-indication to corticosteroids (active gastroduodenal ulcer, uncontrolled sepsis, etc. ..)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
ICU mortality rate | ICU stay (on average patients will be followed 30 days)

SECONDARY OUTCOMES:
Length of MV (and ventilatory free days) | ICU stay (on average patients will be followed 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Fekri Abroug, MD, Principal Investigator — CHU F.Bourguiba Monastir
Locations (1):
- CHU F.Bourguiba, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No
There is no plan to IPD so far

REFERENCES:
- [Background] Chang KC, Leung CC, Kong FY. Corticosteroid administration and treatment failure in acute exacerbation of chronic obstructive pulmonary disease. JAMA. 2010 Oct 13;304(14):1554; author reply 1554-6. doi: 10.1001/jama.2010.1438. No abstract available. PMID 20940378
- [Background] Gunen H, Mirici A, Meral M, Akgun M. Steroids in acute exacerbations of chronic obstructive pulmonary disease: are nebulized and systemic forms comparable? Curr Opin Pulm Med. 2009 Mar;15(2):133-7. doi: 10.1097/MCP.0b013e32832185da. PMID 19532028